CLINICAL TRIAL: NCT01796171
Title: A Phase 1/2 Study of Lutetium (177Lu)-Lilotomab Satetraxetan (Betalutin®) Antibody-radionuclide-conjugate for Treatment of Relapsed Non-Hodgkin Lymphoma.
Brief Title: A Phase 1/2 Study of Betalutin for Treatment of Relapsed Non-Hodgkin Lymphoma
Acronym: LYMRIT-37-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nordic Nanovector (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2011-000033-36
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Results first posted 2024-01-10 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-12

CONDITIONS: Non-Hodgkin Lymphoma; Follicular Lymphoma
Keywords: Radioimmunotherapy; Lu-177; Phase I study; Phase II study; Betalutin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A, Arm 1: 10 MBq/kg Betalutin with lower dose lilotomab pre-dosing (Experimental): 10 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  Interventions: Drug: 10 MBq/kg Betalutin; Drug: 40 mg lilotomab
- Part A, Arm 1: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing (Experimental): 15 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  Interventions: Drug: 15 MBq/kg Betalutin; Drug: 40 mg lilotomab
- Part A, Arm 1: 20 MBq/kg Betalutin with lower dose lilotomab pre-dosing (Experimental): 20 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  Interventions: Drug: 20 MBq/kg Betalutin; Drug: 40 mg lilotomab
- Part A, Arm 2: 10 MBq/kg Betalutin with no pre-dosing (Experimental): 10 MBq/kg (based on body weight) Betalutin without pre-dosing
  Interventions: Drug: 10 MBq/kg Betalutin
- Part A, Arm 2: 15 MBq/kg Betalutin with no pre-dosing (Experimental): 15 MBq/kg (based on body weight) Betalutin without pre-dosing
  Interventions: Drug: 15 MBq/kg Betalutin
- Part A, Arm 3: 15 MBq/kg Betalutin with rituximab pre-dosing (Experimental): 15 MBq/kg (based on body weight) Betalutin with rituximab pre-dosing
  Interventions: Drug: 15 MBq/kg Betalutin; Drug: Rituximab
- Part A, Arm 4: 15 MBq/kg Betalutin with higher dose lilotomab pre-dosing (Experimental): 15 MBq/kg (based on body weight) Betalutin with 100 mg/m2 (based on body surface area) lilotomab pre-dosing
  Interventions: Drug: 15 MBq/kg Betalutin; Drug: 100 mg/m2 lilotomab
- Part A, Arm 4: 20 MBq/kg Betalutin with higher dose lilotomab pre-dosing (Experimental): 20 MBq/kg (based on body weight) Betalutin with 100 mg/m2 (based on body surface area) lilotomab pre-dosing
  Interventions: Drug: 20 MBq/kg Betalutin; Drug: 100 mg/m2 lilotomab
- Part A, Arm 5: 20 MBq/kg Betalutin with intermediate dose lilotomab pre-dosing (Experimental): 20 MBq/kg (based on body weight) Betalutin with 60 mg/m2 (based on body surface area) lilotomab pre-dosing
  Interventions: Drug: 20 MBq/kg Betalutin; Drug: 60 mg/m2 lilotomab
- Part B, Arm 1: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing (Experimental): 15 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  Interventions: Drug: 15 MBq/kg Betalutin; Drug: 40 mg lilotomab
- Part B, Arm 2: 20 MBq/kg Betalutin with higher dose lilotomab pre-dosing (Experimental): 20 MBq/kg (based on body weight) Betalutin with 100 mg/m2 (based on body surface area) lilotomab pre-dosing
  Interventions: Drug: 20 MBq/kg Betalutin; Drug: 100 mg/m2 lilotomab
- Part B, Arm 3: 12.5 MBq/kg Betalutin with lower dose lilotomab pre-dosing (Experimental): 12.5 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  Interventions: Drug: 40 mg lilotomab; Drug: 12.5 mBq/kg Betalutin
- Part C: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing (Experimental): 15 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  Interventions: Drug: 15 MBq/kg Betalutin; Drug: 40 mg lilotomab

INTERVENTIONS:
Drug: 10 MBq/kg Betalutin
  Arms: Part A, Arm 1: 10 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part A, Arm 2: 10 MBq/kg Betalutin with no pre-dosing
Drug: 15 MBq/kg Betalutin
  Arms: Part A, Arm 1: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part A, Arm 2: 15 MBq/kg Betalutin with no pre-dosing; Part A, Arm 3: 15 MBq/kg Betalutin with rituximab pre-dosing; Part A, Arm 4: 15 MBq/kg Betalutin with higher dose lilotomab pre-dosing; Part B, Arm 1: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part C: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing
Drug: 20 MBq/kg Betalutin
  Arms: Part A, Arm 1: 20 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part A, Arm 4: 20 MBq/kg Betalutin with higher dose lilotomab pre-dosing; Part A, Arm 5: 20 MBq/kg Betalutin with intermediate dose lilotomab pre-dosing; Part B, Arm 2: 20 MBq/kg Betalutin with higher dose lilotomab pre-dosing
Drug: 40 mg lilotomab
  Arms: Part A, Arm 1: 10 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part A, Arm 1: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part A, Arm 1: 20 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part B, Arm 1: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part B, Arm 3: 12.5 MBq/kg Betalutin with lower dose lilotomab pre-dosing; Part C: 15 MBq/kg Betalutin with lower dose lilotomab pre-dosing
Drug: 100 mg/m2 lilotomab
  Arms: Part A, Arm 4: 15 MBq/kg Betalutin with higher dose lilotomab pre-dosing; Part A, Arm 4: 20 MBq/kg Betalutin with higher dose lilotomab pre-dosing; Part B, Arm 2: 20 MBq/kg Betalutin with higher dose lilotomab pre-dosing
Drug: 60 mg/m2 lilotomab
  Arms: Part A, Arm 5: 20 MBq/kg Betalutin with intermediate dose lilotomab pre-dosing
Drug: Rituximab
  Arms: Part A, Arm 3: 15 MBq/kg Betalutin with rituximab pre-dosing
Drug: 12.5 mBq/kg Betalutin
  Arms: Part B, Arm 3: 12.5 MBq/kg Betalutin with lower dose lilotomab pre-dosing

SUMMARY:
This study is a Phase 1/2 open-label three part study in patients with relapsed indolent Non-Hodgkin's lymohoma (NHL) (Parts A and C) or relapsed/refractory follicular lymphoma (FL) (Part B).

DETAILED DESCRIPTION:
Part A of the study was a Phase 1/2a study to assess the safety and preliminary efficacy of different treatment regimens of Betalutin with expansion at the candidate recommended Phase 2 doses. Part B was a dedicated Phase 2b randomized substudy to further assess the efficacy and safety of the candidate recommended Phase II doses. Part C was a Phase 2a fixed dose expansion cohort planned to obtain supplementary pharmacokinetic data.

ELIGIBILITY:
Part A and Part C:

Inclusion Criteria:

1. Histologically confirmed (by World Health Organization [WHO] classification) relapsed incurable non-Hodgkin B-cell lymphoma of following subtypes; follicular grade I-IIIA (for Part C, this excludes patients meeting Part B criteria, who should enter Part B), marginal zone, small lymphocytic, lymphoplasmacytic, mantle cell.
2. Age ≥ 18 years.
3. Part A: A pre-study WHO performance status of 0-1; Part C: WHO performance status of 0-2.
4. Life expectancy should be ≥3 months.
5. <25% tumour cells in bone marrow biopsy (biopsy taken from a site not previously irradiated).
6. Measurable disease by radiological methods.
7. Women of childbearing potential must:

   1. understand that the study medication is expected to have teratogenic risk.
   2. have a negative pregnancy test.
   3. agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study medication, throughout study medication therapy and for 12 months after end of study medication therapy, even if she has amenorrhoea.
8. Male patients must agree to use condoms during intercourse throughout study medication therapy and the following 12 months.
9. Patients previously treated with native rituximab are eligible.
10. The patient is willing and able to comply with the protocol, and agrees to return to the hospital for follow up visits and examination.
11. The patient has been fully informed about the study and has signed the informed consent form.

Exclusion Criteria:

Medical contraindications, including uncontrolled infection, severe cardiac, pulmonary, neurologic, psychiatric or metabolic disease, uncontrolled asthma/allergy requiring systemic steroids, known to be human immunodeficiency virus (HIV) positive.

2. Laboratory values within 15 days pre-registration:

1. Absolute neutrophil counts (ANC) ≤1.5×109/L.
2. Part A: Platelet count ≤150×109/L; Part C: Platelet count <150×109/L. For Part C, criteria 2a and 2b must be satisfied within 72 hours of the administration of rituximab
3. Total bilirubin ≥30 mmol/L (Part A only). Total bilirubin > 1.5×ULN (except patients with documented Gilbert's syndrome [≥3.0 mg/dL]) (Part C only).
4. Alkaline phosphatase (ALP) and alanine transaminase (ALT) ≥4×normal level (Part A only).

   Aspartate transaminase (AST), ALT or ALP >2.5×ULN (or >5.0×ULN with liver involvement by primary disease). (Part C only).
5. Creatinine ≥115 µmol/L (men), 97 µmol/L (women) (Part A only). Serum creatinine ≥1.5×ULN (Part C only).
6. Haemoglobin <9.0 g/dL (Part C only). 3. Known central nervous system (CNS) involvement of lymphoma. 4. Previous total body irradiation. 5. Positive test for human anti-murine antibody (HAMA) at screening. 6. Chemotherapy or immunotherapy received within the last 4 weeks prior to start of study treatment. Pre treatment with rituximab is allowed.

   7. Pregnant or lactating women. 8. Previous hematopoietic stem cell transplantation (autologous and allogenic). 9. Part A: Previous treatment with radioimmunotherapy. Part C: Not applicable. 10. Actively participating in another study or received an IMP within 4 weeks prior to enrolment.

   11. Receipt of live-attenuated vaccine within 30 days prior to enrolment. 12. Part A and Part C: Test positive for hepatitis B (HBsAg and anti-HBc). Part C only: Test positive for hepatitis C and human immunodeficiency virus (HIV).

   13. A known hypersensitivity to rituximab, lilotomab, Betalutin or murine proteins or any excipient used in rituximab, lilotomab, or Betalutin.

   Part B:

   Inclusion Criteria:

   Histologically confirmed (by WHO classification) relapsed non-Hodgkin B-cell FL (grade I IIIA).

   2. Male or female aged ≥18 years. 3. Received at least 2 prior systemic anti-neoplastic or immunotherapy-based regimens (maintenance therapy following a CR/PR is not considered to be a separate line of therapy). Systemic regimens including agents such as idelalisib or other PI3K inhibitors qualify as a prior line of therapy.

   4. Prior therapy must have included a rituximab/anti-CD20 agent and an alkylating agent - which may be been administered in separate regimens.

   5. Patients must be refractory to any at least one previous regimen that contained rituximab or an anti CD20 agent, with refractoriness defined as:

i. no response (no CR or PR) during therapy, or ii. a response (CR/PR) lasting less than 6 months after the completion of a regimen including rituximab/anti-CD20 therapy (including occurrence of progressive disease (PD) during rituximab/anti-CD20 maintenance therapy, or within 6 months of completion of maintenance therapy).

6. WHO performance status of 0-2. 7. Life expectancy of ≥3 months. 8. Bone marrow tumour infiltration <25% (in biopsy taken from a site not previously irradiated).

9. Measurable disease by CT or MRI: longest diameter (LDi) >1.5 cm for nodal lesion, LDi >1.0 cm for extra nodal lesion on an assessment performed during the screening period.

Criteria 10 and 11 must be satisfied within 72 hours of the administration of rituximab:

10. ANC ≥1.5×109/L. 11. Platelet count ≥100×109/L.

Criteria 12 to 15 must be verified at time of eligibility review within 2 weeks prior to rituximab administration:

12. Haemoglobin ≥9.0 g/dL. 13. Total bilirubin ≤1.5×upper limit of normal (ULN) (except patients with documented Gilbert's syndrome [<3.0 mg/dL]).

14. Liver enzymes: AST; ALT or ALP ≤2.5×ULN (or ≤5.0×ULN with liver involvement by primary disease).

15. Adequate renal function as demonstrated by a serum creatinine <1.5×ULN. 16. Women of childbearing potential must:

1. understand that the study medication is expected to have teratogenic risk.
2. have a negative serum beta human-chorionic gonadotropin (ß-HCG) pregnancy test at screening.
3. commit to continued abstinence from heterosexual intercourse (excluding periodic abstinence or the withdrawal method) or begin a highly effective method of birth control with a Pearl-Index <1%, without interruption, from 4 weeks before starting study medication, throughout study medication therapy and for 12 months after end of study medication therapy, even if she has amenorrhoea. Apart from abstinence, highly effective methods of birth control are: i. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).

ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) iii. Intrauterine device (IUD). iv. Intrauterine hormone-releasing system (IUS). v. Bilateral tubal occlusion. vi. Vasectomised partner. 17. Male patients must agree to use condoms during intercourse throughout study treatment administration and for 12 months following administration of Betalutin.

18. The patient is willing and able to comply with the protocol, and agrees to return to the hospital for follow up visits and examination.

19. The patient has been fully informed about the study and has signed the informed consent form.

20. Negative HAMA test at screening. 21. Negative test at screening for Hepatitis B (negative HBsAg and anti-HBc), Hepatitis C and HIV.

Exclusion Criteria

1. Prior hematopoietic allogenic stem cell transplantation.
2. Patients with a prior autologous SCT are excluded unless at least two years have elapsed since transplantation.
3. Evidence of histological transformation from FL to diffuse large B-cell lymphoma (DLBCL) at time of screening (transformation to grade IIIB that was successfully treated with recurrence of grade I-IIIA initial clone is accepted).
4. Previous total body irradiation.
5. Prior anti-lymphoma therapy (chemotherapy, immunotherapy or other systemic agent including any investigational agent) within 4 weeks prior to start of study treatment (corticosteroid treatment at doses of ≤ 20 mg/day, topical or inhaled corticosteroids, granulocyte colony-stimulating factor [G-CSF] or granulocyte-macrophage colony-stimulating factor [GM-CSF] are permitted up to 2 weeks prior to start of rituximab)..
6. Patients who are receiving any other investigational medicinal products.
7. Patients with known or suspected CNS involvement of lymphoma.
8. History of malignancy other than FL within 5 years prior to screening( i.e. patients with cancer diagnosed within 5 years prior to screening or who were diagnosed prior to 5 years and were not in CR or were on treatment within 5 years prior to screening), with the exception of malignancies with a negligible risk of metastasis or death (e.g. 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localised prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.

.9. Pregnant or breastfeeding women. 10. Exposure to another CD37 targeting drug. 11. A known hypersensitivity to rituximab, lilotomab, Betalutin or murine proteins or any excipient used in rituximab, lilotomab, or Betalutin.

12. Has received a live-attenuated vaccine within 30 days prior to enrolment. 13. Evidence of severe or uncontrolled systemic diseases:

1. Uncontrolled infection including evidence of ongoing systemic bacterial, fungal, or viral infection (excluding viral upper respiratory tract infections) at the time of initiation of study treatment.
2. Pulmonary conditions e.g. unstable or uncompensated respiratory disease.
3. Hepatic, renal, neurological, or metabolic conditions - which in the opinion of the investigator would compromise the protocol objectives.
4. Psychiatric conditions e.g. patients unlikely to comply with the protocol, e.g. mental condition rendering the patient unable to understand the nature, scope, and possible consequences of participating in the study.
5. History of erythema multiforme, toxic epidermal necrolysis, or Stevens-Johnson syndrome.
6. Cardiac conditions in the previous 24 weeks (before date of consent), including

i. history of acute coronary syndromes (including unstable angina). ii. class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.

iii. known uncontrolled arrhythmias (except sinus arrhythmia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Freitag, Study Director — Nordic Nanovector
Locations (96):
- United States (14):
  - University Of Arkansas For Medical Sciences, Little Rock, Arkansas
  - Pacific Shores Medical Group, Long Beach, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Dallas, Texas
- Royal Hobart Hospital, Hobart, Australia
- Austria (2):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Medizinische Universität Wien - AKH Wien, Universitaetsklinik fuer Innere Medizin I, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Gent (UZ Gent), Ghent
  - CH Jolimont, La Louvière
  - UZ Leuven, Leuven
- Canada (3):
  - London Health Sciences Centre, London
  - Sault Area Hospital, Sault Ste. Marie
  - Princes Margaret Cancer Centre, Toronto
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (2):
  - University Hospital Olomouc, Olomouc
  - FNsP Ostrava, Ostrava-Poruba
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Odense Univerisity Hospital, Odense
- Finland (2):
  - Helsinki University Hospital Comprehensive Cancer Center, Helsinki
  - Central Hospital Of Central Finland, Jyväskylä
- France (6):
  - Institut Bergonie, Bordeaux
  - Chu Grenoble - Hopital Michallon, Grenoble
  - Hôpital Saint Louis, Paris
  - AP-HP La Pitié salpétrière, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Regional Universitaire de Tours (CHRU de Tours) - Hopital Bretonneau, Tours
- Hungary (2):
  - Orszagos Onkologiai Intezet, A-Belgyogyaszati Onkologiai Osztaly, Budapest
  - Semmelweis Egyetem, I Belgyogyaszati Klinika, Hematologiai Osztaly, Budapest
- Ireland (3):
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (6):
  - Haemek Medical Center, Afula
  - Asaf Harofeh Medical Center, Be’er Ya‘aqov
  - Bnai Zion Medical Center (BZMC), Haifa
  - Rambam Health Care Campus (RHCC), Haifa
  - יHadassah Ein Karem Medical Center, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Italy (8):
  - SS Antonio & Biagio and C. Arrigo Hospital, Alessandria
  - "Istituto di Ematologia ed Oncologia Medica "" L. & A. Seragnoli""-Policlinico S. Orsola Malpighi", Bologna
  - Universita Degli Studi Di Firenze-Azienda Ospedaliero-Universitaria Careggi (AOUC), Florence
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola
  - Istituto Europeo di Oncologia (IEO), Milan
  - "Istituto Nazionale Tumori Fondazione G. Pascale", Napoli
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - AO Ordine Mauriziano di Torino, Torino
- University Medical Center Groningen, Groningen, Netherlands
- Norway (3):
  - Haukeland Universitetssjukehus, Bergen
  - The Norwegian Radium Hospital, Oslo
  - St Olav Hospital, Trondheim
- Poland (3):
  - Szpital Morski Im.Pck W Gdynia, Gdynia
  - Pratia MCM Kraków, Krakow
  - Centrum Onkologii, Warsaw
- National University Hospital, Singapore, Singapore
- South Korea (3):
  - Chonbuk National University Hospital, Jeonju
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (9):
  - Corporacio Sanitaria Parc Taulí, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Clinica Universidad De Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Health Research Institute La Fe - Hospital La Fe, Valencia
  - Hospital Universitario Doctor Peset, Valencia
- Cancercentrum -Center of Oncology, Umeå, Sweden
- Kantonsspital Graubünden, Chur, Switzerland
- Turkey (Türkiye) (10):
  - Cukurova Universitesi Tip Fakültesi, Ic Hastaliklari Anabilim Dali, Adana
  - Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi Ic, Ankara
  - Hacettepe University Oncology Hospital, Ankara
  - Eskisehir Osmangazi Universitesi Tip Fakultesi Ic Hastaliklar, Eskişehir
  - Istanbul Universitesi Istanbul Tip Fakultesi, Fatih
  - Ege Universitesi Tip Fakültesi, Izmir
  - Celal Bayar Universitesi Tip Fakultesi, Manisa
  - Ondokuz Mayis Universitesi, Samsun
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama, Şehitkamil
- United Kingdom (9):
  - Dorset Cancer Centre Poole Hospital, Poole, Dorset
  - Bristol Haematology and Oncology Centre, Bristol
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - University College London Hospitals Nhs Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Derriford Hospital, Plymouth
  - The Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Background] Dahle J, Repetto-Llamazares AH, Mollatt CS, Melhus KB, Bruland OS, Kolstad A, Larsen RH. Evaluating antigen targeting and anti-tumor activity of a new anti-CD37 radioimmunoconjugate against non-Hodgkin's lymphoma. Anticancer Res. 2013 Jan;33(1):85-95. PMID 23267131
- [Background] Repetto-Llamazares AH, Larsen RH, Mollatt C, Lassmann M, Dahle J. Biodistribution and dosimetry of (177)Lu-tetulomab, a new radioimmunoconjugate for treatment of non-Hodgkin lymphoma. Curr Radiopharm. 2013 Mar;6(1):20-7. doi: 10.2174/1874471011306010004. PMID 23256748
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Derived] Londalen A, Blakkisrud J, Revheim ME, Madsbu UE, Dahle J, Kolstad A, Stokke C. FDG PET/CT parameters and correlations with tumor-absorbed doses in a phase 1 trial of 177Lu-lilotomab satetraxetan for treatment of relapsed non-Hodgkin lymphoma. Eur J Nucl Med Mol Imaging. 2021 Jun;48(6):1902-1914. doi: 10.1007/s00259-020-05098-x. Epub 2020 Nov 16. PMID 33196921
- [Derived] Kolstad A, Illidge T, Bolstad N, Spetalen S, Madsbu U, Stokke C, Blakkisrud J, Londalen A, O'Rourke N, Beasley M, Jurczak W, Fagerli UM, Kascak M, Bayne M, Obr A, Dahle J, Rojkjaer L, Pascal V, Holte H. Phase 1/2a study of 177Lu-lilotomab satetraxetan in relapsed/refractory indolent non-Hodgkin lymphoma. Blood Adv. 2020 Sep 8;4(17):4091-4101. doi: 10.1182/bloodadvances.2020002583. PMID 32877524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the Australia, Canada, the European Union, Israel, Norway, Singapore, Turkey, United Kingdom (UK) and United States (US)
Pre-assignment Details: 255 patients were screened in the 28 days before the start of treatment, 191 were enrolled, 190 started pre-treatment with rituximab (one enrolled participant died before starting rituximab) and 187 were treated with Betalutin
Groups:
- Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 10 MBq/kg Betalutin
  40 mg lilotomab
- Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 15 MBq/kg Betalutin
  40 mg lilotomab
- Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 20 MBq/kg Betalutin
  40 mg lilotomab
- Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing: 10 MBq/kg Betalutin
- Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing: 15 MBq/kg Betalutin
- Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing: 15 MBq/kg Betalutin
  Rituximab
- Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing: 15 MBq/kg Betalutin
  100 mg/m2 lilotomab
- Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing; Part B, Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing: 20 MBq/kg Betalutin
  100 mg/m2 lilotomab
- Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing: 20 MBq/kg Betalutin
  60 mg/m2 lilotomab
- Part A Received Rituximab Only; Part B Received Rituximab Only: Did not receive pre-dosing or Betalutin
- Part B, Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 15 MBq/kg Betalutin
  40 mg lilotomab
  These two groups were combined for analysis and reporting as they were run in parallel and participants received the same treatment
- Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 40 mg lilotomab
  12.5 mBq/kg Betalutin
- Enrolled But Not Treated: Participants were enrolled but did not receive any study treatment
Period: Enrolled
Arm/Group | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing | Part A Received Rituximab Only | Part B, Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B, Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B Received Rituximab Only | Enrolled But Not Treated
Started | 4 | 36 | 3 | 1 | 2 | 3 | 3 | 18 | 4 | 2 | 76 | 28 | 9 | 1 | 1
Completed | 4 | 36 | 3 | 1 | 2 | 3 | 3 | 18 | 4 | 2 | 76 | 28 | 9 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Pre-reatment With Rituximab
Arm/Group | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing | Part A Received Rituximab Only | Part B, Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B, Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B Received Rituximab Only | Enrolled But Not Treated
Started (Started pre-treatment with rituximab) | 4 | 36 | 3 | 1 | 2 | 3 | 3 | 18 | 4 | 2 | 76 | 28 | 9 | 1 | 0
Completed | 4 | 36 | 3 | 1 | 2 | 3 | 3 | 18 | 4 | 0 | 76 | 28 | 9 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Period With Betalutin
Arm/Group | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing | Part A Received Rituximab Only | Part B, Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B, Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B Received Rituximab Only | Enrolled But Not Treated
Started | 4 | 36 | 3 | 1 | 2 | 3 | 3 | 18 | 4 | 0 | 76 | 28 | 9 | 0 | 0
Completed | 4 | 35 | 3 | 1 | 2 | 3 | 3 | 18 | 3 | 0 | 65 | 25 | 8 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 11 | 3 | 1 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Start of further anticancer therapy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing | Part A Received Rituximab Only | Part B, Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B, Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B Received Rituximab Only | Enrolled But Not Treated
Started | 4 | 35 | 3 | 1 | 2 | 3 | 3 | 18 | 3 | 0 | 65 | 25 | 8 | 0 | 0
Completed | 0 | 5 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 30 | 2 | 1 | 2 | 3 | 2 | 18 | 2 | 0 | 65 | 25 | 8 | 0 | 0
Not completed — Start of further anticancer therapy | 4 | 25 | 2 | 1 | 2 | 2 | 1 | 15 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 17 | 9 | 1 | 0 | 0
Not completed — Patient transferred to other hospital | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 40 | 15 | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants receiving rituximab
Groups:
- Part A - Received Rituximab Only; Part B - Received Rituximab Only: Participant received pre-treatment only and was withdrawn before receiving Betalutin
- Part B Arm 1 and Part and C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 15 MBq/kg Betalutin
  40 mg lilotomab
  Note: these two groups were combined for the purposes of the safety analyses as they received the same treatment therefore have been combined for the purposes of reporting baseline variables for consistency
- Total: Total of all reporting groups
Arm/Group | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing | Part A - Received Rituximab Only | Part B Arm 1 and Part and C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B, Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B - Received Rituximab Only | Total
Number analyzed (Participants) | 4 | 36 | 3 | 1 | 2 | 3 | 3 | 19 | 3 | 2 | 76 | 28 | 9 | 1 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 11 | 1 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 29 | 9 | 4 | 1 | 63
  >=65 years | 2 | 25 | 2 | 1 | 2 | 3 | 2 | 15 | 2 | 2 | 47 | 19 | 5 | 0 | 127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 19 | 0 | 0 | 1 | 2 | 0 | 9 | 1 | 2 | 46 | 16 | 3 | 1 | 101
  Male | 3 | 17 | 3 | 1 | 1 | 1 | 3 | 10 | 2 | 0 | 30 | 12 | 6 | 0 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 36 | 3 | 1 | 2 | 3 | 3 | 19 | 3 | 2 | 73 | 23 | 9 | 1 | 182
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Part A, Phase I
Description: Number of participants with dose limiting toxicities (DLTs) in Part A
Time Frame: 12 weeks
Population: Population evaluable for DLTs. Note one further participant was treated with 20 MBq Betalutin and 100 mg/m2 lilotomab but was underdosed with lilotomab so was not evaluable for DLTs and has not been included.
Measure: Count of Participants; unit: Participants
Groups:
- Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 10 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  10 MBq/kg Betalutin
  40 mg lilotomab
- Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 15 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  15 MBq/kg Betalutin
  40 mg lilotomab
- Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 20 MBq/kg (based on body weight) Betalutin with 40 mg lilotomab pre-dosing
  20 MBq/kg Betalutin
  40 mg lilotomab
- Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing: 15 MBq/kg (based on body weight) Betalutin with rituximab pre-dosing
  15 MBq/kg Betalutin
  Rituximab
- Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing: 15 MBq/kg (based on body weight) Betalutin with 100 mg/m2 (based on body surface area) lilotomab pre-dosing
  15 MBq/kg Betalutin
  100 mg/m2 lilotomab
- Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing: 20 MBq/kg (based on body weight) Betalutin with 100 mg/m2 (based on body surface area) lilotomab pre-dosing
  20 MBq/kg Betalutin
  100 mg/m2 lilotomab
- Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing: 20 MBq/kg (based on body weight) Betalutin with 60 mg/m2 (based on body surface area) lilotomab pre-dosing
  20 MBq/kg Betalutin
  60 mg/m2 lilotomab
Arm/Group | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing
Number analyzed (Participants) | 4 | 6 | 3 | 1 | 2 | 3 | 3 | 6 | 3
Participants | 0 | 1 | 3 | 0 | 2 | 1 | 1 | 1 | 0

2. Primary Outcome: Part A, Phase IIa
Description: Tumour response rates in patients in Part A receiving Betalutin based on evaluation of CT scan images including PET/CT imaging (and bone marrow biopsy if applicable).
Time Frame: 5 years
Population: Per-protocol analysis set: participants receiving Betalutin who had adequate tumour assessments at baseline, and after ≥12 weeks (unless disease progression occurred), and no major protocol deviations impacting on efficacy results. Only participants in Phase IIa with FL receiving 40/15 and 100/20 With FL were analyzed. This was the analysis set selected for efficacy analysis as this was the population selected for further analysis in the larger Part B study.
Measure: Count of Participants; unit: Participants
Groups:
- 40/15 With FL: Participants in the PPS in Phase IIa with follicular lymphoma who received 15 MBq/kg Betalutin and 40 mg lilotomab
- 100/20 With FL: Participants in the PPS in Phase IIa with follicular lymphoma who received 20 MBq/kg Betalutin and 100 mg/m2 lilotomab
Arm/Group | 40/15 With FL | 100/20 With FL
Number analyzed (Participants) | 18 | 9
Participants
  Complete remission | 7 | 2
  Partial remission | 5 | 6
  Stable disease | 3 | 1
  Progressive disease | 3 | 0

3. Primary Outcome: Part B, Phase IIb
Description: Overall response rate in Part B defined as the number of participants with a best response of complete remission or partial remission at any time
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- 40/15 in Part B: Participants in Part B with FL who received 40 mg lilotomab and 15 MBq/kg Betalutin
- 100/20 in Part B: Participants in Part B with FL who received 100 mg/m2 lilotomab and 20 MBq/kg Betalutin
- 40/12.5 in Part B: Participants in Part B with FL who received 40 mg lilotomab and 12.5 MBq/kg Betalutin
Arm/Group | 40/15 in Part B | 100/20 in Part B | 40/12.5 in Part B
Number analyzed (Participants) | 72 | 28 | 9
Participants | 28 | 9 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from informed consent up to 12 weeks after Betalutin administration (note: in Part A SAEs only were collected between informed consent and rituximab administration; in Parts B and C all adverse events were collected in this period). Treatment-related adverse events were then collected up to 5 years (end of the study).
Description: Summaries of adverse events were generated for all participants
Groups:
- Part A Rituximab Only; Part B Rituximab Only: Did not receive pre-dosing or Betalutin
- Part B Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 15 MBq/kg Betalutin
  40 mg lilotomab
  These two groups were combined for analysis and reporting as they were run in parallel and participants received the same treatment
- Part B Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing: 20 MBq/kg Betalutin
  100 mg/m2 lilotomab
- Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing: 12.5 mBq/kg Betalutin
  40 mg lilotomab
- Part B Not Treated: Enrolled but died before receiving rituximab
Arm/Group | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing | Part A Rituximab Only | Part B Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing | Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing | Part B Rituximab Only | Part B Not Treated
All-Cause Mortality (participants affected / at risk) | 2/4 | 10/36 | 0/3 | 0/1 | 0/2 | 2/3 | 2/3 | 6/18 | 1/4 | 0/2 | 23/76 | 11/28 | 1/9 | 0/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 7/36 | 2/3 | 0/1 | 2/2 | 1/3 | 1/3 | 0/18 | 0/4 | 0/0 | 12/76 | 7/28 | 0/9 | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 3/4 | 36/36 | 3/3 | 0/1 | 2/2 | 3/3 | 3/3 | 16/18 | 4/4 | 2/2 | 61/76 | 22/28 | 9/9 | 1/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=4) | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=36) | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=3) | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing (N=1) | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing (N=2) | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing (N=3) | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing (N=3) | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing (N=18) | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing (N=4) | Part A Rituximab Only (N=0) | Part B Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=76) | Part B Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing (N=28) | Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=9) | Part B Rituximab Only (N=1) | Part B Not Treated (N=1)
Chronic myelomonocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 1 | 0 | 0 | NA
Pharygngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 2 | 1 | 0 | 0 | NA
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 2 | 0 | 0 | 0 | NA
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0 | 0 | 0 | NA
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Pleural infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 1 | 0 | 0 | NA
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 1 | 0 | 0 | NA
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
squamous cell carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 2 | 0 | 0 | 0 | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 1 | 0 | 0 | NA
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 1 | 0 | 0 | NA
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 1 | 0 | 0 | NA
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0 | 0 | 0 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | NA
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | 1 | 0 | NA | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | NA | 0 | 0 | 0 | NA | NA | NA | 0 | 0 | NA | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Arm 1: 10 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=4) | Part A, Arm 1: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=36) | Part A, Arm 1: 20 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=3) | Part A, Arm 2: 10 MBq/kg Betalutin With no Pre-dosing (N=1) | Part A, Arm 2: 15 MBq/kg Betalutin With no Pre-dosing (N=2) | Part A, Arm 3: 15 MBq/kg Betalutin With Rituximab Pre-dosing (N=3) | Part A, Arm 4: 15 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing (N=3) | Part A, Arm 4: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing (N=18) | Part A, Arm 5: 20 MBq/kg Betalutin With Intermediate Dose Lilotomab Pre-dosing (N=4) | Part A Rituximab Only (N=2) | Part B Arm 1 and Part C: 15 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=76) | Part B Arm 2: 20 MBq/kg Betalutin With Higher Dose Lilotomab Pre-dosing (N=28) | Part B, Arm 3: 12.5 MBq/kg Betalutin With Lower Dose Lilotomab Pre-dosing (N=9) | Part B Rituximab Only (N=1) | Part B Not Treated (N=1)
Neutropenia (Blood and lymphatic system disorders) | 2 | 20 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 12 | 3 | 3 | 0 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 19 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 13 | 3 | 3 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 14 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 10 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 2 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 12 | 6 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 5 | 3 | 0 | 2 | 3 | 2 | 3 | 2 | 0 | 2 | 2 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 3 | 3 | 0 | 1 | 3 | 2 | 3 | 1 | 0 | 6 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 4 | 2 | 0 | 1 | 2 | 1 | 4 | 0 | 0 | 8 | 3 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 3 | 0 | 0 | 1 | 1 | 4 | 1 | 0 | 3 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Blood lactate dehydrogenase decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 10 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 8 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 11 | 3 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 5 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 4 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Hypermobility syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Rash macropapular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetitie (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dose calculation error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Percussion test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (4):
  • Study Protocol (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT01796171/Prot_000.pdf
  • Statistical Analysis Plan: Part A main SAP (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT01796171/SAP_001.pdf
  • Statistical Analysis Plan: Part A SAP addendum (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT01796171/SAP_002.pdf
  • Statistical Analysis Plan: Part B and C SAP (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT01796171/SAP_003.pdf